CLINICAL TRIAL: NCT03962725
Title: Eliminating Use of Non Depolarizing Neuromuscular Blocking Agents to Reduce Postoperative Pulmonary Complications: A Multi-center, Randomized Control Trial
Brief Title: Avoiding Neuromuscular Blockers to Reduce Complications
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study terminated due to lack of enrollment.
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Maximilian S Schaefer, Assistant Professor of Anaesthesia, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2019P000260
Record Dates: First submitted 2019-05-21; First posted 2019-05-24 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Respiratory Failure; Respiratory Infection; Aspiration Pneumonia; Pneumonitis; Atelectasis; Bronchospasm
Keywords: Neuromuscular Blocker Avoidance; Post Operative Pulmonary Complications; General Anesthesia Maintenance; Inhaled Anesthetics
MeSH Terms: conditions — Respiratory Insufficiency; Respiratory Tract Infections; Pneumonia, Aspiration; Pneumonia; Pulmonary Atelectasis; Bronchial Spasm | interventions — Neuromuscular Blocking Agents; Rocuronium; Analgesics, Opioid; Propofol; Dexmedetomidine; Ketamine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group (C) (Active Comparator): Endotracheal intubation would be facilitated by either Rocuronium (0.6-1mg kg-1) or Succinylcholine (1-1.5mg kg-1) and further dosing of Rocuronium would be left at the discretion of the anesthesia team members. Choice and technique of induction and maintenance of anesthesia, use of vasopressors, perioperative antibiotics, analgesics/adjunct regional techniques, prophylaxis for postoperative nausea and vomiting, fluid and blood component therapy would be left at the discretion of the anesthesia team. Neuromuscular blockade would be reversed with either Sugammadex or Neostigmine (based on institutional availability) and trachea would be extubated once patient meets criteria per attending anesthesiologist.
  Interventions: Drug: Neuromuscular Blocking Agents
- No Relaxant Group (NR) (Experimental): Endotracheal intubation would be facilitated by Succinylcholine (1-1.5mg/kg) or Remifentanil (1-2mcg kg-1) if Succinylcholine use is contraindicated. No non-depolarizing NMBA would be administered to the patients randomized to the NR group. Choice and technique of induction and maintenance of anesthesia, use of vasopressors, perioperative antibiotics, analgesics/adjunct regional techniques, prophylaxis for postoperative nausea and vomiting, fluid and blood component therapy would be left at the discretion of the anesthesia team. Use of deeper plane of inhaled anesthetics or adjuncts (opioids, propofol, dexmedetomidine or ketamine) either as boluses or infusion would be recommended in case of sustained high peak airway pressures (>35mm Hg), high intra-abdominal pressure, involuntary patient/diaphragmatic movement hindering surgical exposure and dissection. Choice and dose of adjunct/s to optimize operating conditions would be left to the discretion of the anesthesia team.
  Interventions: Drug: Anesthetic Adjuncts

INTERVENTIONS:
Drug: Neuromuscular Blocking Agents — Use of non depolarizing neuromuscular blocking agents for maintenance of general anesthesia.
  Other Names: Rocuronium
  Arms: Control Group (C)
Drug: Anesthetic Adjuncts — Use of deeper plane of inhaled anesthetics or adjuncts (opioids, propofol, dexmedetomidine or ketamine for maintenance of general anesthesia.
  Other Names: opioids, propofol, dexmedetomidine or ketamine
  Arms: No Relaxant Group (NR)

SUMMARY:
The goal of this study to evaluate whether eliminating the use of non-depolarizing neuromuscular blocking agents (NMBA) for maintenance of general anesthesia reduces postoperative pulmonary complications in higher risk patients.

DETAILED DESCRIPTION:
Pragmatic prospective randomized controlled assessor-blinded effect-size finding trial involving approximately 100 patients total at two academic tertiary care hospitals: Beth Israel Deaconess Medical Center (BIDMC) and Massachusetts General Hospital (MGH). Patients will be randomized into one of two study groups: standard care group which uses Rocuronium (NMBA) as an adjunct for maintenance of general anesthesia and non-relaxant arm that avoids the use of NMBA and instead uses additional inhalational anesthetics, opioids, propofol, dexmedetomidine, or ketamine for maintenance of general anesthesia. Assessment of postoperative pulmonary complications and in-hospital mortality would be achieved by close review of the patient's medical records during the hospital stay, for a maximum of 28 days.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Undergoing non-cardiac surgery under general anesthesia with an endotracheal tube
* those at higher risk of developing postoperative pulmonary complications (internally validated risk prediction score of >=20)

Exclusion Criteria:

* Emergency surgery
* Ambulatory (outpatient) surgery
* Scheduled for elective postoperative ventilation
* Planned return to operating room within 7 days of index procedure
* Exposure to general anesthesia within 7 days prior to planned procedure
* Requirement mechanical ventilation at baseline (not including stable use of CPAP/BiPAP)
* Pregnant patients: as detected by patient self-reporting or diagnosed by preoperative pregnancy testing according to institutional policies at BIDMC and MGH
* Allergy to either non-depolarizing muscle relaxants or sugammadex
* Clinician refusal
* Prisoner

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2019-08-07 (Actual); Primary Completion 2022-12-19 (Actual); Study Completion 2022-12-19 (Actual)

PRIMARY OUTCOMES:
Number of participants who either had postoperative pulmonary complications or died in hospital within 28 days of index procedure. | 28 Days
  Composite of respiratory failure, suspected respiratory infection, aspiration pneumonia or pneumonitis, atelectasis, bronchospasm, reintubation and all cause in-hospital mortality

SECONDARY OUTCOMES:
Vasopressor Use Between Groups | During the surgery
  Vasopressor equivalent dose
Duration of Intraoperative Hypotension | During the surgery
  Mean arterial pressure <55mmHg
Surgeon's Assessment of surgical field | During the surgery
  Was the operative condition optimal for the surgeon graded qualitatively using a numerical rating scale of 1-4. A score of 1 indicates excellent operating conditions whereas 4 indicates conditions unacceptable to the surgeon.

OTHER OUTCOMES:
30-Day Readmission Rates | 30 days
  How often patients had to be readmitted to the hospital within 30 days of discharge from hospital following index procedure.
Time to Post-Anesthesia Care Unit (PACU) Discharge Readiness | Day after surgery
  Time is takes for patients to be ready for discharge from PACU post operatively.
Cost of Anesthetic Medication | During the surgery
  Cost of anesthetics used during surgical procedures in the study.
Rate of Unplanned ICU Admission or Return to Operating Room | 24 hours
  How often patients had either unanticipated ICU admissions or return to the operating room within 24 hours of the initial operation.
Hospital Length of Stay | Upto 30 days
  How much total time patients spent in the hospital after the operation.

CONTACTS AND LOCATIONS:
Overall Officials: Maximilian S Schaefer, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No